CLINICAL TRIAL: NCT04250168
Title: Piloting Clinical Bacteriology in the Ebola Virus Disease Care Response to Detect Intercurring Bloodstream Infections and Inform Appropriate Antibiotic Treatment
Brief Title: Piloting Clinical Bacteriology in the Ebola Virus Disease Care Response
Acronym: Bact_EVD
Status: Terminated | Type: Observational
Why Stopped: Ebola epidemic in N-Kivu has ended
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other); Alliance for International Medical Action (Other); Médecins Sans Frontières, France (Other); International Medical Corps (Unknown); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 1328/19
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-02

CONDITIONS: Sepsis Bacterial; Ebola Virus Disease; Bloodstream Infection
Keywords: Ebola Virus Disease; EVD; Bacterial infections; bacteriology; blood cultures; CRP; DR Congo; Antibiotic Resistance; Bacterial bloodstream infection
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Sepsis; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite access to experimental Ebola Virus Disease (EVD)-specific treatments, about 30% of patients still die in the Ebola Treatment Centers (ETC) in DRC. There is limited study done about the potential contribution of bacterial co-infections (in particular bloodstream infections) to this adverse outcome, as blood cultures were so far rarely available in epidemic areas. Findings from patients treated in Europe and the USA, and case discussions in the field call for further investigation.

Building further on an ongoing microbiological surveillance project of ITM and INRB in DRC, we are able to set up a research project which will pilot in a standardized manner clinical bacteriology tools (bacterial blood cultures, biomarkers as CRP, procalcitonin and white blood cell differential count, and clinical early warning scores) to study bacterial bloodstream infection in EVD patients in the N-Kivu/Ituri outbreak.

This project will add evidence on 1) frequency, causative pathogen and antibiotic resistance profiles of bacterial bloodstream infections, as well as 2) the predictive value of biomarkers and early warning scores, in EVD patients at different timepoints during hospitalization in an ETC in DRC. The results will inform appropriate antibiotic treatment in an EVD setting and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted in an Ebola Treatment Center (ETC) or Ebola Transit Center (TC)
* Laboratory-confirmed (Ebola RT-PCR positive result) EVD diagnosis, or, EVD suspect patient requiring instant intravenous antibiotic treatment
* Willing and able to provide written informed consent personally or by a legally acceptable representative if the patient is unable to do so

Exclusion Criteria:

* We do not exclude certain patient groups, but whenever harm is expected from the additional blood sampling needed for this study, the clinician can opt not to enroll the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of laboratory confirmed EVD patients admitted to the Ebola Treatment Centers (ETCs) in N-Kivu & Ituri province and participating in the study. As broad-spectrum antibiotics are often started as soon as patients arrive in the suspect area of the ETC or transit center, and as this might interfere with bacterial bloodstream infection detection in blood cultures, patients can be included from the stage of being 'a probable suspect' onwards in some instances (i.e. prior to start-up of broad-spectrum antibiotics, clinical suspicion of bacterial bloodstream infection at admission in suspect area, etc).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Determine frequency, causative pathogen, and antibiotic resistance profiles of bacterial bloodstream infections among confirmed EVD patients | 7 months
  Proportion of patients with grown blood cultures versus those who were sampled, spectrum of bacterial species and proportion of antibiotic resistance

SECONDARY OUTCOMES:
Assess the value of simple biomarker blood tests (WBC + DIFF, CRP, PCT) and Early Warning Scores (EWS) to guide targeted empiric antibiotic treatment and to early detect bacterial bloodstream infections, as compared to bacterial blood culture results | 7 months
  Relation between score and or biomarker level and growth from blood cultures
Validate current empiric antibiotic treatment guidelines in EVD care | 7 months
  Proportion of cases for which empiric antibiotic covered the bacteria causing bloodstream infections

CONTACTS AND LOCATIONS:
Overall Officials: Octavia Lunguya, Principal Investigator — INRB; Jan Jacobs, Principal Investigator — ITM
Locations (2):
- Democratic Republic of the Congo (2):
  - Ebola Treatment Centers, Beni/Mangina, N-Kivu/Ituri
  - institut national de recherche biomedicale(INRB), Kinshasa